CLINICAL TRIAL: NCT03547648
Title: Comparison of the Effect of Three Different Peak Airway Pressures on Determining Intraoperative Bleeding Points in Thyroidectomies
Brief Title: Effect of Three Different Peak Airway Pressures on Determining Intraoperative Bleeding in Thryroidectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, Anaesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 172208
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Thyroid Neoplasms; Thyroid Nodule
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I ( 30 cm H2O) (Active Comparator): Patients will be applied 30 cm H2O peak airway pressure manually at the end of the surgery
  Interventions: Procedure: peak airway pressure
- Group II( 40 cm H2O) (Active Comparator): Patients will be applied 40 cm H2O peak airway pressure manually at the end of the surgery
  Interventions: Procedure: peak airway pressure
- Group III(50 cm H2O) (Active Comparator): Patients will be applied 50 cm H2O peak airway pressure manually at the end of the surgery
  Interventions: Procedure: peak airway pressure

INTERVENTIONS:
Procedure: peak airway pressure — Patients' peak airway pressures will be raised to observe intraoperative bleeding in thyroidectomy surgery. Aim is to prevent postoperative bleeding.

SUMMARY:
Patients undergoing thyroidectomy will be divided into three groups (30 cm H2O Group I, 40 cm H2O Group II, 50 cmH2O Group III). At the end of the operation patients will be applied peak airway pressure manually according to involved groups.The time until the first hemorrhage is seen in each group or if not seen pressure will be applied for 30 seconds and then will be ended.We will record the blood pressure, spO2, HR, the first ETCO2 after the procedure, postoperative haemorrhage that required surgery, and postoperative hematomas during peak airway pressure increase during the operation in all patients. The 1st hour blood pressure, nausea-vomiting score and pain score (NRS) will be recorded in the postoperative recovery unit.

The primary end point of the study is intraoperative bleeding detected, and the secondary end point is postoperative bleeding.

DETAILED DESCRIPTION:
Patients will be divided into three groups (https://www.randomizer.org/) by computer assisted randomization method (30 cm H2O in Group I, 40 cm H2O in Group II, 50 cmH2O in Group III peak pressure will be applied). The time until the first hemorrhage is seen in each group or if not seen pressure will be applied for 30 seconds and then will be ended.

Patients will be taken to the operation table and standard monitorization will be performed consisting of ECG, non-invasive blood pressure and peripheral O2 saturation from the back region. Anesthesia was induced with 2 mg / kg propofol (propofol 1% Fresenius, Fresenius Kabi, Germany), 2 mg / kg fentanyl (Talinat 0,5mg / 10ml, AND, Turkey), 0.6 mg / kg rocuronium (Muscuro 50mg / 5ml, Kocak Farma , Turkey) will be provided after the patients were intubated orally. General anesthesia treatment will be provided with 2% Sevoflurane in 40% oxygen-air mixture. All patients will be ventilated in pressure controlled mode; respiratory frequency: 12 / min, FiO2: 40% (oxygen-air mixture), I/E:1/2, PEEP: 7 cmH2O supplying end tidal CO2 value of 32-36 mmHg.

Calculating the ideal weight of the patient, isolated-S (Polifarma, Turkey)2ml/kg/h will be infused. If the systolic arterial pressure (SAB) or heart rate (HR) increases by 20% compared to baseline, IV 50 μg fentanyl will be administered. At the end of the operation, the patient's airway peak pressure will be increased before hemostasis is provided by the same surgeon (S.T.). Positive pressure on the Maquet Flow I device (Maquet Flow I-AGC, Rastatt, USA) will be applied manually(30 cm H2O in Group I, 40 cm H2O in Group II patients and 50 cm H2O in group III patients). The airway peak pressure increase will be maintained and recorded until the surgeon sees the first bleeding point or if not seen for 30 seconds. For all three groups this process will be repeated one more time.

After peak airway pressure is increased, the number of bleeding centers detected, how long time did it take to detect and the size of the bleeding vessel (<2 mm or> 2 mm)will be recorded. We will record the blood pressure, spO2, HR, the first ETCO2 after the procedure, postoperative haemorrhage that required surgery, and postoperative hematomas during peak airway pressure increase during the operation in all patients. The 1st hour blood pressure, nausea-vomiting score and pain score (NRS) will be recorded in the postoperative recovery unit.

The primary end point of the study is intraoperative bleeding detected, and w the secondary end point is postoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II patients
* Patients undergoing total thyroidectomy
* Aged between 18-60 years

Exclusion Criteria:

* Active pulmonary disease
* Cardiac aritmia
* Intracranial mass
* Coagulation defects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding point | 30 seconds
  Determination of intraoperative bleeding point just after applying positive airway pressure manually

SECONDARY OUTCOMES:
postoperative haemorrhage | 24 hours
  Postoperative haemorrhage for 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akcivan, resident, Study Chair — Istanbul University; Aylin Özdilek, MD, Study Chair — Istanbul University; Emre Erbabacan, Ass Prof, Study Chair — Istanbul University; Fatiş Altındaş, Prof, Study Chair — Istanbul University; Serkan Teksöz, Ass Prof, Study Chair — Istanbul University
Locations (1):
- Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar CM, Van Zundert AAJ. Intraoperative Valsalva maneuver: a narrative review. Can J Anaesth. 2018 May;65(5):578-585. doi: 10.1007/s12630-018-1074-6. Epub 2018 Jan 24. PMID 29368315
- [Result] Tokac M, Dumlu EG, Bozkurt B, Ocal H, Aydin C, Yalcin A, Cakir B, Kilic M. Effect of Intraoperative Valsalva Maneuver Application on Bleeding Point Detection and Postoperative Drainage After Thyroidectomy Surgeries. Int Surg. 2015 Jun;100(6):994-8. doi: 10.9738/INTSURG-D-15-00002.1. PMID 26414819
- [Derived] Beyoglu CA, Teksoz S, Ozdilek A, Akcivan M, Erbabacan E, Altindas F, Koksal G. A comparison of the efficacy of three different peak airway pressures on intraoperative bleeding point detection in patients undergoing thyroidectomy: a randomized, controlled, clinical trial. BMC Surg. 2020 Apr 10;20(1):69. doi: 10.1186/s12893-020-00728-5. PMID 32276609